CLINICAL TRIAL: NCT04634305
Title: Evaluation of the Clinical and Functional Results Obtained After a Total Elbow Arthroplasty, All Indications Combined
Brief Title: Clinical and Functional Results After Total Elbow Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, François SIRVEAUX, Clinical Professor François Sirveaux, Central Hospital, Nancy, France
Other Study IDs: 2020PI204
Record Dates: First submitted 2020-10-18; First posted 2020-11-18 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Elbow Fracture; Elbow Arthropathy; Elbow Osteoarthritis
MeSH Terms: conditions — Elbow Fractures | interventions — Arthroplasty, Replacement, Elbow

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 72 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Total elbow arthroplasty: Total elbow arthroplasty, all indications combined
  Interventions: Procedure: Total elbow arthroplasty

INTERVENTIONS:
Procedure: Total elbow arthroplasty — Total elbow arthroplasty by a single operator

SUMMARY:
Analysis of clinical and functional outcomes after a total elbow arthrosplasty, all indications combined, with a minimum follow up of 24 months The hypothesis is that there a significant improvement after an elbow replacement, no matter what the surgery indication is

ELIGIBILITY:
Inclusion Criteria:

* Total elbow arthroplasty, all indication combined

Exclusion Criteria:

* Less than 24 months of follow up
* Revision of total elbow arthroplasty

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Every patient that underwent a total elbow arthroplasty between january 2004 and august 2020 by a single operator in our orthopedic center
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2004-01-01 (Actual); Primary Completion 2006-02-01 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Mayo Elbow Performance Score | through study completion, an average of 5 years
QuickDASH | through study completion, an average of 5 years
Range of motion | through study completion, an average of 5 years

SECONDARY OUTCOMES:
Implant loosening | through study completion, an average of 5 years
  Radiolucent lines around the implant on the X Ray
Triceps deficiency | through study completion, an average of 5 years
Bushing wear | through study completion, an average of 5 years
  Measure of an angle on the X Ray

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: Undecided